CLINICAL TRIAL: NCT00611273
Title: A Multi-center Long Term Efficacy Trial of the GFX For Reduction of Glabellar Furrowing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advanced Cosmetic Intervention (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACI 007-02; WIRB 20062119
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Glabellar Furrowing
Keywords: Glabellar Furrowing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients who have presented to the investigator for correction of glabellar furrows, as classified per the Rated Numeric Kinetic Line Scale Score for Facial Wrinkles Secondary to Hyperkinetic Function (Note: Class 1 or Higher)7 (Appendix R) are candidates for this study.
  Interventions: Device: GFX

INTERVENTIONS:
Device: GFX — The GFX system employs minimally invasive technique utilizing Bi-polar (radio frequency) RF technology. GFX ablates nerves activating the muscles that cause glabellar furrowing.
  Other Names: RF Nerve Ablation Device

SUMMARY:
Long term efficacy study of GFX for patients undergoing reduction of glabellar furrowing

DETAILED DESCRIPTION:
A Multi-center Long Term Efficacy Trial of GFX for the Reduction of Glabellar Furrowing

ELIGIBILITY:
Inclusion Criteria: The patient will be included if:

* Has no medical contraindication
* Presents for correction of glabellar furrows, as classified per the Rated Numeric Kinetic Line Scale Score for Facial Wrinkles Secondary to Hyperkinetic Function (Class 1 or Higher)
* Is at least 18 years of age
* Signs a written informed consent
* Understands and accepts the obligation to present for scheduled follow-up visits
* Understands that the GFX procedure may not be successful
* Presents at the one month follow-up visit with an improvement from the base line RNKLS score

Exclusion Criteria: The patient will be excluded if:

* Has had an injection of botulinum toxin to the target area within the previous 4 months and still exhibits a positive cosmetic effect to the glabellar frown.
* Has had silicone, fat, collagen or a synthetic material placed in the glabellar region or surgical correction or excision of the glabellar furrows
* Has a known bleeding disorder
* Pregnant
* Has received or is anticipated to receive anti-platelets, anti-coagulants, thrombolytics, or cancer therapy
* Is receiving systemic corticosteroids or anabolic steroids (standard doses of inhaled or nasal corticosteroids are acceptable)
* Has a history of chronic or recurrent infection or compromised immune system
* Has severe allergies manifested by a history of anaphylaxis
* Has known lidocaine hypersensitivity
* Is enrolled in another study
* Has history of keloid formation
* The investigator believes the patient is not a suitable candidate for the GFX procedure, or is not likely to receive cosmetic benefitPresents at the one month follow-up visit with no improvement from the base line RNKLS score

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Time at which the patient no longer shows an improvement from the base line RNKLS score indicating that the initially successful GFX procedure is no longer effective at a scheduled follow-up visit. | 18 months

SECONDARY OUTCOMES:
Minimal or transient incidence of minor unanticipated adverse events. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: James Newman, MD, Study Director — Premier Plastic Surgery
Locations (10):
- United States (9):
  - Paul S. Nassif, MD, FACS, Beverly Hills, California
  - James Newman, San Mateo, California
  - Michael E. Jansin, MD, Tampa, Florida
  - Foad Nahai, M.D., F.A.C.S., Atlanta, Georgia
  - Steven P. Block, MD, Highland Park, Illinois
  - Keith LaFerriere, MD, Springfield, Missouri
  - J. Smythe Rich, III, M.D, Columbia, South Carolina
  - Russell W. Kridel, MD, Houston, Texas
  - Roger C. Mixter, MD, Milwaukee, Wisconsin
- David A. Ellis, MD, Toronto, Ontario, Canada